CLINICAL TRIAL: NCT03759704
Title: Investigating Metabolic Characteristics of Musculoskeletal Sarcoma In Vivo Using Hyperpolarized Carbon-13 Magnetic Resonance Spectroscopic Imaging (MRSI)
Brief Title: Metabolic Characteristics of Sarcoma In Vivo Using HP 13-C Magnetic Resonance Spectroscopic Imaging (MRSI)
Acronym: HPMSS
Status: Withdrawn | Type: Observational
Why Stopped: No participants meeting inclusion criteria were found.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jae Mo Park, Principal Investigator, University of Texas Southwestern Medical Center
Other Study IDs: STU 072017-069
Record Dates: First submitted 2018-04-11; First posted 2018-11-30 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Musculoskeletal Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperpolarized 13CPyruvate and gadolinium: Injection with hyperpolarized 13CPyruvate followed by gadolinium during MRSI.
  Interventions: Drug: Hyperpolarized 13CPyruvate

INTERVENTIONS:
Drug: Hyperpolarized 13CPyruvate — Bolus injection of study drug during MRSI.
  Other Names: HP Pyruvate injection

SUMMARY:
Investigators will determine whether MRSI using hyperpolarized [1-13C]pyruvate provide useful information of tumor malignancy in MRI-indeterminate cases. Metabolite maps of hyperpolarized [1-13C]lactate and H13CO3- produced from hyperpolarized [1-13C]pyruvate will be compared to the biopsy results of MRI-indeterminate patients and the 13C-maps of age-matched healthy subjects.

DETAILED DESCRIPTION:
A non-randomized, interventional (nontherapeutic), feasibility trial to detect metabolic changes in participants with musculoskeletal sarcoma using hyperpolarized [1-13C]pyruvate Magnetic Resonance Spectroscopy Imaging (MRSI). All measured quantities will be tabulated and the analysis will be descriptive and obervational in nature.

Participants in this study will receive the study drug, hyperpolarized [1-13C]pyruvate, as a bolus injection during an MRSI of either a soft tissue sarcoma or healthy tissue. After the study drug injection and MRSI, participants will then receive contrast material, Gadavist, via injection during continuation the MRI.

ELIGIBILITY:
Inclusion Criteria:

SARCOMA patients:

- MRI indeterminate solid enhancing lesion in the pelvis or extremity.

ALL subjects:

* Age 18 through 100 years.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.
* All races and ethnicities will be included; subjects must be able to read and speak the English or Spanish language.

Exclusion Criteria:

SARCOMA patients:

-Subjects who have had radiotherapy to the indeterminate lesion.

ALL subjects:

* Subjects who have had chemotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Subjects may not be receiving any other investigational agents.
* Any contraindication per MRI Screening form including implants contraindicated at 3T, pacemakers, implantable Cardioverter Defibrillator (ICD), claustrophobia.
* Metallic foreign bodies in the field of view which may interfere with MRI acquisitions.
* Since each subject is receiving a gadolinium based contrast agent intravenously, additional contraindications would include: eGFR ≤ 30 mL/min/1.73m2, sickle cell disease, or hemolytic anemia.
* Uncontrolled psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible study participants will be identified by referring physicians from a UT Southwestern Clinic. A treating physician will discuss the potential research opportunity with their patient to determine interest in study participation.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
The product ratio difference of lactate to bicarbonate in tumor bearing regions from those in the normal-appearing tissue. | One day visit with injection during MRSI
  How much metabolic contrast can be detected using hyperpolarized Carbon-13 pyruvate

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Imaging Research Center, Dallas, Texas, United States